CLINICAL TRIAL: NCT00774865
Title: Long Term Follow-up of Robotic Assisted Surgical Revascularization With CT Angiography
Brief Title: Long Term Follow-up of Robotic Assisted Surgical Revascularization
Acronym: ZEUSFUPCTA
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: R-08-190; 15000
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
Keywords: Robotic; CABG; LITA; Patency; Long; Term
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical: Patients who have previously undergone robotic bypass surgery
  Interventions: Procedure: MIBI and CTA

INTERVENTIONS:
Procedure: MIBI and CTA — Rest and Stress MIBI and CT Angiography

SUMMARY:
The objectives of the 2-year study are two-fold:

1. To determine the 5-7 year patency rate (rate of open bypass grafts) of the LITA graft of patients who have already had robotically-assisted CABG surgery using CTA and MPS-MIBI
2. To determine patient quality of life at 5-7 years after robotically-assisted CABG surgery

DETAILED DESCRIPTION:
New techniques such as robotically-assisted CABG surgery need proper evaluation to ensure potential benefits gained are not harmful to that which we know to be of significant benefit to the patients, that being the left internal thoracic artery (LITA) graft (one of the main coronary arteries supplying your heart with blood). We are therefore proposing a 5-7 year CT-Angiography (CTA) and Myocardial Perfusion Scintigraphy (MPS-MIBI) to assess the patency rate of the LITA graft in patients that have already undergone robotically assisted CABG.

Between September 1999 and December 2001, a single surgeon performed robotically-assisted CABG surgery with LITA-to-LAD anastomosis on 151 patients with single vessel coronary artery disease at the London Health Sciences Centre, University Hospital. Patient consent and Research Ethics approval from The University of Western Ontario was acquired prior to each procedure. Sixty-one patients had robotically-assisted CABG surgery using the Automated Endoscopic Stabilizer for Optimal Positioning (AESOP) 3000 (Computer Motion, Goleta, CA), while 90 patients had robotically-assisted CABG surgery using the Zeus telemanipulation surgical system (Computer Motion, Goleta, CA). The AESOP 3000 is a single-arm robot that facilitates video thoracoscopic LITA dissection by providing steady images and voice-activated camera control. The Zeus telemanipulation surgical system is a multi-arm robotic telemanipulator that incorporates AESOP and allows control of surgical instruments within the thorax from a distant console.

Postoperative angiography was completed prior to discharge whenever possible. Patients continue to be followed on an annual basis. Our intent to perform follow-up angiography and MPS-MIBI at 5 and 10 years duration to assess LITA graft performance was discussed with each patient at the time of the original surgery. Two late deaths unrelated to surgery have been recorded in this cohort.

The 2-year study will be divided into three phases: Phase I - Patient Recruitment (4 months), Phase II - Patient Assessment with CTA, MPS-MIBI and Questionnaires (16 months) and Phase III - Data Analysis and Conclusions (4 months).

Phase I - Chart Review and Patient Recruitment (4 Months) Upon receiving approval from the Research Ethics Board at The University of Western Ontario, charts will be reviewed on all 151 robotically-assisted CABG surgery patients. Data on these patients is currently stored in a regularly updated database at our institution; however, a thorough review of all charts will be performed. Patient demographics and operative notes, as well as perioperative and postoperative complications will be reviewed. Hospital admissions, documented cardiac events and any subsequent deaths not previously documented will be recorded. Any additional pertinent data from the chart review will be entered into a study specific Microsoft Excel file maintained by a single qualified research assistant.

All 149 living robotically-assisted CABG surgery patients will be contacted and their participation in the study requested. Patients will receive an initial request by mail, with an informative letter signed by the principal investigator outlining the purpose of the study, what participation in the study involves, and the specific aims of the cardiac team at the conclusion of the study. A follow-up phone call will be done within 3-weeks of mailing the letter to go over the content and answer any questions that patients may have.

Phase II - Patient Assessment via CTA, MPS-MIBI and Questionnaires (16 Months)

Robotically-assisted CABG surgery patients that agree to be a part of the study will have arrangements made for them to travel to LHSC. Patients will undergo a structured half-day (approximately 4-6 hours) at the hospital consisting of the following:

1. Selective coronary artery and LITA graft check via CTA with a 64 slice CT scanner + Rest MPS-MIBI then Stress MPS-MIBI (4-6hrs)
2. Completion of two validated health related quality of life questionnaires

   1. Seattle Angina Questionnaire
   2. 36-Item Short Form Health Survey

ELIGIBILITY:
Inclusion Criteria:

1. Have had previous robotically-assisted CABG surgery with a LITA to LAD anastomosis with either AESOP or Zeus performed between September 1999 and December 2001 at the London Health Sciences Centre
2. Willing to give informed consent to participate in the study

Exclusion Criteria:

1. Expired
2. Unable or unwilling to give informed consent
3. History of allergic reaction to contrast material used in CTA or severe adverse reactions to medications used in MPS-MIBI procedures

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All 150 living robotically-assisted CABG surgery patients will be contacted and their participation in the study requested. Patients will receive an initial request by mail, with an informative letter signed by the principal investigator outlining the purpose of the study, what participation in the study involves, and the specific aims of the cardiac team at the conclusion of the study. A follow-up phone call will be done within 3-weeks of mailing the letter to go over the content and answer any questions that patients may have.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine the 5-7 year patency rate of the LITA graft of patients who have already had robotically-assisted CABG surgery using CTA and MPS-MIBI | 5-7 years post robotic assisted CABG

SECONDARY OUTCOMES:
To determine patient quality of life at 5-7 years after robotically-assisted CABG surgery | 5-7 years post robotic assisted CABG

CONTACTS AND LOCATIONS:
Overall Officials: Bob Kiaii, MD, FRCSC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada